CLINICAL TRIAL: NCT00363935
Title: A Randomized, Double-blind, Controlled Study of Dexmedetomidine (Precedex) Infusion for Improving Control of Acute Autonomic Response During Laparoscopic Bariatric Surgery
Brief Title: Bariatric Dose-ranging Study With Dexmedetomidine
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 072005-020
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Abdominal Surgery Patients
MeSH Terms: interventions — Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine

SUMMARY:
After obtaining informed consent,80 morbidly obese ASA II-III patients undergoing laparoscopic bariatric surgery procedures would be randomly assigned to one of four study groups at UTSWMC at Dallas.Hemodynamic paarameters, recovery times, postoperative pain scores, the need for rescue analgesics and side effects will be recorded.The purpose of this study is to determine the optimal linfusion rate of dexmedetomidine for maintaining cardiovscular stability during general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included in the study only if they meet all of the following criteria:

1. Age 18 to 70 years
2. Undergo laparoscopic bariatric surgery requiring general anesthesia
3. Be capable of giving informed consent
4. ASA physical status I-III ( Appendix 1)

Exclusion Criteria:

1. Subjects will be excluded from the study for any of the following reasons:
2. With history of hypertension and allergy to dexmedetomidine
3. Patients who have greater than first degree heart block.
4. Performing major intracavitary surgery procedures
5. Patients who are pregnant or breast-feeding
6. History of alcohol or drug abuse

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01-01 (Estimated); Primary Completion 2007-01-01 (Estimated); Study Completion 2007-01-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Paul White, MD, PhD, Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- The University of Texas Southwestern MedicalCenter at Dallas, Dallas, Texas, United States